CLINICAL TRIAL: NCT04169243
Title: Randomized Controlled Trial Intervention With New Nordic DIet in Women With GestatiOnal Diabetes Mellitus: iNDIGO
Acronym: iNDIGO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Post-pandemic women did not engage in unnecessary tasks. Changes were made (more languages and sites, short proof-of-concept study, easier recepies, food for whole family, social media, etc. After 4 yr 5 women were recruited and trial terminated
Sponsor: Göteborg University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iNDIGO2018-00483
Record Dates: First submitted 2019-10-28; First posted 2019-11-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome is percentage of time in target of blood glucose values, measured with continuous glucose monitoring. The device will be masked for participants. Still, because the trial is a diet intervention, participants will know their group status. However, initial data reaching the Investigators will not have the code broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Women randomized to the New Nordic Diet meet the study dietician at week 30 for 1.5 hr of individual diet treatment according to the New Nordic Diet and a cognitive behavioral approach. The diet advice include evenly distributed meals over the day, foods low in fat and rich in fibre, 500 g fruit and vegetables daily, fish 2-3 times a week and keyhole foods. Participants will prepare their own food but are provided with recipes and food bags containing ingredients and foods to be consumed during the two-week intervention At gestational age 32 weeks, women meet with a dietitian and will be instructed to continue with the New Nordic Diet diet throughout pregnancy on their own.
  Interventions: Behavioral: New Nordic Diet
- Control (Active Comparator): The control women receive diet advice according to usual care.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: New Nordic Diet — The New Nordic Diet conforms with the Nordic Nutrition Recommendations and incorporates environmental sustainability and planetary health. It includes rapeseed oil, whole grain bread, wild fish, seafood and game, potatoes, root vegetables, cabbages, Nordic fruits and berries. A two-week menu including all daily meals has been created to ensure dietary goals of the New Nordic Diet intervention: fish and shellfish intake ≥ 3 times/w (fatty fish at least once per week), ≥ 500 g fruit, berries, vegetables and legumes daily (legumes as main protein source at least twice per week), whole-grain cereal products, rapeseed oil for cooking/dressing and three table spoons of nuts and seeds per day.
  Arms: Intervention
Other: Control — The control women receive diet advice according to usual care, which may be a short meeting with the regular midwife or a short meeting with a dietician. From the study, they will receive a gift certificate that can be used in grocery stores.
  Arms: Control

SUMMARY:
The study evaluates whether the New Nordic Diet, compared to routine care, will improve glucose control, among women developing gestational diabetes mellitus during pregnancy.

Originally, a 10 wk intervention with qualified counseling on New Nordic Diet was planned, and effects on glycosylated haemoglobin A (HbA1c) at gestational age 37 weeks was planned as main outcome. Recruitment started in spring 2020 but had to be halted due to covid-19. Instead, we now conduct a more comprehensive version of the study, with a more intensive intervention consisting of distributed food bags plus dietary counselling for two weeks, and with continuous glucose monitoring during these two weeks to measure main outcome. This is more sensitive to small changes than is HbA1c. With this shorter and more intensive intervention we believe we can address our original hypothesis yet adjust to impacts of the covid-19 situation on the population and health care system.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is associated with severe adverse outcomes for mother and newborn. Recently introduced Swedish guidelines on GDM diagnosis will at least double the prevalence of diagnosed women. The first line of treatment in GDM is diet and exercise treatment. Even so, there is a recognized knowledge gap as to what diet treatment is optimal. In routine care today, diagnosed women are provided by midwife with the same diet advice as patients with diabetes type 2 and these are broad and general. Only rarely are the diet advice provided by a dietician. In nutrition research, most evidence for health benefits of a diet has been demonstrated for the Mediterranean diet. Further, the New Nordic Diet (NND) was recently developed to mimic the Mediterranean diet yet builds on foods grown in the Nordic climate, thus focusing on gastronomical potential and sustainability. Interestingly, a diet intake in line with NND among Norwegian mothers was associated with lower risk for excessive pregnancy weight gain. In addition, associations have been shown between NND and lower risk for cardiovascular disease, obesity, inflammatory risk markers, serum lipids, colorectal cancer and total mortality. Hence, it seems likely that diet treatment with NND to women with GDM would be superior to routine care, but this has never been investigated. The main aim of the randomized controlled trial Intervention with new Nordic DIet in women with GestatiOnal diabetes mellitus (iNDIGO) is to test if the NND compared with usual care will improve glucose control in women with GDM. The iNDIGO study is a randomized parallel, single-blinded, controlled trial. In total, 50 women diagnosed with GDM are recruited and randomized to receive either a NND (intervention) or usual care (control) for 14 days. Participants receive a two-week menu and provided with food bags containing ingredients for dishes and foods to be used. Primary outcome is glycemic control (specifically time in target) measured using continuous glucose monitoring. Compliance to the dietary intervention will be tested using known dietary biomarkers and adherence questionnaires. Maternal socio-demographic and clinical data, biological samples, dietary intake and physical activity will be collected at enrollment and at the end of intervention (30-32 weeks' gestation).

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with diagnosis of gestational diabetes in pregnancy wks 24-28.

Exclusion Criteria:

* multiple pregnancies
* not understanding/able to read Swedish or English
* unwilling to follow a dietary intervention
* manifest diabetes

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Time in Target at gestational week 32 | At week 32 of pregnancy
  Percentage of time in target (TIT) range 3.5-7.8 mmol/L measured with continuous glucose monitoring

SECONDARY OUTCOMES:
Pregnancy weight gain | Pre-pregnant weight up to delivery
  Weight gain during pregnancy from self-reported pre-pregnancy weight until delivery
Incidence of pregnancy-induced hypertension | Up to delivery
  Diagnosis of pregnancy-induced hypertension
Incidence of pre-eclampsia | Up to delivery
  Diagnosis of pre-eclampsia
Prevalence of use of insulin/Metformin treatment | Up to delivery
  Decision to put woman on medication for the gestational diabetes, such as metformin or insulin
Incidence of preterm delivery | Up to 37 completed weeks
  Delivery before 37 completed weeks
Incidence of Caesarean sections | Up to delivery
  Delivery by caesarean sections
Health-related quality of life | Up to 1 year postpartum
  Health-related quality of life, calculated from questionnaire information from RAND-36
Incidence of LGA | At delivery
  Large-for-gestational age born infant
Incidence of shoulder displacement | At delivery
  Shoulder displacement of newborn infant
Apgar scores measurements | At delivery
  Apgar scores measured at 1, 5 and 10 minutes after delivery
Additional measurements from continuous glucose monitoring at wk 32 | At gestational week 32
  mean glucose, CV, SD, MAGE, % time with values >7.8 mmol/L, % time with values <3.5 mmol/L, glucose in different time periods, and AUC
Additional measurements from continuous glucose monitoring at wk 36 | At gestational week 36
  mean glucose, CV, SD, MAGE, % time with values >7.8 mmol/L, % time with values <3.5 mmol/L, glucose in different time periods, and AUC
Incidence of macrosomia | At delivery
  Diagnosis of macrosomia in newborn infant
Nutritional status | During pregnancy
  Nutritional status (vitamins and minerals) of mother during pregnancy
Diet quality measuremen¨t | Up to delivery
  Diet intake quality of mother during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Anna Winkvist, PhD, Principal Investigator — Göteborg University
Locations (3):
- Sweden (3):
  - Antenatal care, Gothenburg
  - Region Stockholm, Stockholm
  - Region Västerbotten, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karlsson T, Augustin H, Lindqvist M, Otten J, Petersson K, Storck-Lindholm E, Mogren I, Winkvist A. Effect of the New Nordic Diet compared with usual care on glucose control in gestational diabetes mellitus: Study protocol for the randomized controlled trial intervention with new Nordic DIet in women with GestatiOnal diabetes mellitus (iNDIGO). Contemp Clin Trials. 2022 Apr;115:106706. doi: 10.1016/j.cct.2022.106706. Epub 2022 Feb 12. PMID 35158086